CLINICAL TRIAL: NCT04191148
Title: A Multi-Center Randomized, Double-Blind Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LBP-EC01 in Patients With Lower Urinary Tract Colonization Caused by E. Coli
Brief Title: Safety, Tolerability, and PK of LBP-EC01 in Patients With Lower Urinary Tract Colonization Caused by E. Coli
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Locus Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: LBx-1001
Record Dates: First submitted 2019-12-04; First posted 2019-12-09 (Actual); Results first posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2021-11

CONDITIONS: Urinary Tract Infections
Keywords: UTI; Bacteriophage; Phage
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: 2:1 randomized, placebo controlled, blinded study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LBP-EC01 (Experimental): crPhage cocktail
  Interventions: Drug: LBP-EC01
- Placebo (Placebo Comparator): Lactated Ringer's solution, injection, USP
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LBP-EC01 — crPhage cocktail: at approximately 1.5 x 10^10 to 3.0 x 10^10 PFU/vial dosed BID by intraurethral administration
  Arms: LBP-EC01
Drug: Placebo — Lactated Ringers Solution for Injection dosed BID by intraurethral administration
  Arms: Placebo

SUMMARY:
Study LBx-1001 is a multi-center randomized, double-blind study to assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of LBP-EC01 in patients with indwelling urinary catheters, or requiring intermittent catheterization, and/or patients with asymptomatic bacteriuria caused by Escherichia coli (E. coli). This study population has been selected because LBP-EC01 is a phage cocktail where active bacterial host engagement is required to allow for amplification of the phage and evaluation of the safety and PK of the phage cocktail. Eligible patients will require confirmation of colonization with a urine sample taken within 10 days of randomization that cultures contain ≥10^3 E. coli colony forming unit (CFU)/mL, without the patient having clinical signs or symptoms of an active urinary tract infection (UTI) requiring antibiotic treatment. Patients should have E. coli as the primary colonizing bacteria and must not have a secondary bacterial colonization at levels equal to or greater than that seen from E. coli.

DETAILED DESCRIPTION:
Approximately 30 patients 18 years of age or older with a history of urinary tract infection or colonization caused by E. coli who have indwelling urinary catheters, or who require intermittent catheterization, and/or patients with asymptomatic bacteriuria caused by E. coli colonization (≥10^3 CFU/mL) on microbiological diagnosis, without clinical signs or symptoms of infection requiring antibiotic treatment will be enrolled. Patients will be screened for presence of E. coli colonization (≥10^3 CFU/mL) prior to randomization and evaluated for potential bacterial susceptibility to LBP-EC01.

Secondary Objective: To evaluate the pharmacodynamics (PD) of LBP-EC01. Exploratory Objective: To explore the influence of LBP-EC01 on the urinary tract microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Males or females 18 years of age or older.
4. Patients with a lower urinary tract colonization caused by E. coli (≥10^3 CFU/mL) and who meet at least one of the following criteria:

   * Has an indwelling urinary catheter and medical documentation of a urinary tract infection by E. coli within the past 12 months
   * Requires intermittent catheterization and medical documentation of a urinary tract infection by E. coli within the past 12 months
   * Has medical documentation of a history of asymptomatic bacteriuria (i.e., lower urinary tract colonization) with E. coli at least once in the past 12 months
5. Patients must have experience with urinary catheterization or have Medical Monitor approval if the patient does not have prior experience with catheterization.
6. In good general health as evidenced by medical history and physical examination.
7. Women of childbearing potential and men with female partners of childbearing potential must use two forms of effective contraception, at least 1 of which is a physical barrier method, during the study and which is recommended to continue for 2 weeks after completing the study.

Exclusion Criteria:

1. Patients with clinical signs of active UTI or other infection requiring antimicrobial treatment. These may include dysuria, urinary frequency, urinary urgency, suprapubic discomfort and flank pain in addition to non-specific symptoms of urinary leakage, change in voiding habits, worsening muscle spasm, increasing autonomic dysreflexia, sweating, malaise, and fever or hypothermia. Analgesic use is permitted.
2. Patients who have received Gram-negative bacteria antimicrobials within 14 days of randomization.

   Note: Patients who are currently only receiving antibiotics with only Gram-positive activity (e.g., vancomycin, daptomycin, linezolid) to treat active infections against Gram-positive non-UTIs can be included in the trial.
3. Presence of a surgically-modified bladder, except for a repaired ruptured bladder.
4. History of severe autonomic dysreflexia, which is defined as those patients who have a spinal cord injury and who have had a documented sudden increase in systolic blood pressure of greater than 40 mm Hg due to an irritation or stimulation (including bladder or bowel irritation) below the level of the spinal cord injury. Autonomic dysreflexia can include findings of hypertensive crisis or emergency, clinically significant bradycardia/tachycardia, severe headache or other severe reaction requiring an acute intervention, so consultation with the Medical Monitor should take place if a history of severe autonomic dysreflexia is suspected but not clearly identified.
5. Active severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, or neurologic disease per the investigator's discretion.
6. Any malignancies within the past 5 years (except those in remission).
7. Unless deemed acceptable by the Investigator, prescription drugs, over-the-counter (OTC) medications and supplements that acidify the urine are excluded.
8. Patients who have had allergic reactions to similar compounds, or any excipients.
9. Participation in an investigational drug or device study within 1 month (or 7 half-lives of drug, whichever is longer) prior to randomization.
10. Patients who are pregnant or expecting to conceive, are breast feeding or are planning to breast feed, within 1 month of completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Pinnacle Research Group, Anniston, Alabama
  - Tilda Research, Irvine, California
  - Universal Axon Clinical Research, Doral, Florida
  - Universal Axon - Homestead, LL, Homestead, Florida
  - AMPM Research Clinic, Miami Gardens, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina

REFERENCES:
- [Derived] Lenneman BR, Fernbach J, Loessner MJ, Lu TK, Kilcher S. Enhancing phage therapy through synthetic biology and genome engineering. Curr Opin Biotechnol. 2021 Apr;68:151-159. doi: 10.1016/j.copbio.2020.11.003. Epub 2020 Dec 10. PMID 33310655

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Lactated Ringer's solution injection dosed BID by intraurethral administration
Period: Overall Study
Arm/Group | LBP-EC01 | Placebo
Started | 24 | 12
Completed | 22 | 12
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- LBP-EC01: crPhage cocktail
  LBP-EC01: crPhage cocktail
- Placebo: Lactated Ringer's solution, injection, USP
  Lactated Ringers Solution for Injection: Placebo
- Total: Total of all reporting groups
Arm/Group | LBP-EC01 | Placebo | Total
Number analyzed (Participants) | 24 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (16.36) | 70.5 (14.37) | 67.9 (15.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 10 | 31
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 14 | 4 | 18
  Unknown or Not Reported | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 22 | 11 | 33
  Race: Black or African American | 1 | 1 | 2
  Race: American Indian or Alaska native | 0 | 0 | 0
  Race: Asian | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Other | 1 | 0 | 1
Baseline height (cm) [Mean (Standard Deviation); unit: centimeters] — Population: 2 participants in the experimental group (LBP-EC01) discontinued treatment early
  centimeters
    number analyzed (Participants) | 22 | 12 | 34
    (all) | 162.4 (8.94) | 164.9 (8.86) | 163.3 (8.86)
Baseline weight (kg) [Mean (Standard Deviation); unit: kilograms] — Population: 2 participants in the experimental group (LBP-EC01) discontinued treatment early
  kilograms
    number analyzed (Participants) | 22 | 12 | 34
    (all) | 79.39 (16.555) | 73.04 (9.446) | 77.15 (14.616)
Baseline body mass index (kg/m^2) [Mean (Standard Deviation); unit: kilograms per meters squared] — Population: 2 participants in the control group (LBP-EC01) discontinued treatment early
  kilograms per meters squared
    number analyzed (Participants) | 22 | 12 | 34
    (all) | 30.14 (5.908) | 26.90 (3.280) | 28.99 (5.316)
Frequency of prior UTI in the last 12 months, n(%) [Count of Participants; unit: Participants]
  0 | 10 | 8 | 18
  1 | 12 | 2 | 14
  > 1 | 2 | 2 | 4
Frequency of prior UTI in last 1 month, n(%) [Count of Participants; unit: Participants]
  0 | 12 | 10 | 22
  1 | 11 | 2 | 13
  > 1 | 1 | 0 | 1
Prior antibiotic use (within 30 days of Screening), n(%) [Count of Participants; unit: Participants]
  Yes | 4 | 0 | 4
  No | 20 | 12 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by DAIDS v2.1
Description: Safety and tolerability of LBP-EC01: Number of participants with treatment-related adverse events as assessed by DAIDS v2.1
Time Frame: 35 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | LBP-EC01 | Placebo
Number analyzed (Participants) | 24 | 12
Participants | 0 | 0

2. Primary Outcome: Pharmacokinetics of LBP-EC01: Cmax
Description: Maximum concentration determined directly from the concentration-time profile
Time Frame: 28 days
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: PFU/mL
Arm/Group | LBP-EC01
Number analyzed (Participants) | 24
PFU/mL | 4600000 (37000)

3. Primary Outcome: Pharmacokinetics of LBP-EC01: Tmax
Description: Time to maximum concentration
Time Frame: 28 days
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | LBP-EC01
Number analyzed (Participants) | 24
hours | 2.19 (127.32)

4. Primary Outcome: Pharmacokinetics of LBP-EC01: AUC
Description: Area under the concentration versus time curve from time 0 to the last measurable concentration
Time Frame: 28 days
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*PFU/ mL
Arm/Group | LBP-EC01
Number analyzed (Participants) | 24
h*PFU/ mL | 13000000 (69000)

5. Secondary Outcome: Reduction in Urinary E.Coli Burden at Any of the Following Time Points: Day 2, Day 3, Day 5, Day 7 (EOT), Day 14 and Day 28
Description: The secondary objective of this study was to evaluate the pharmacodynamics (PD) of LBP-EC01 through reduction in urinary E.coli burden as defined by at least 1 log CFU reduction from baseline.
Time Frame: 28 days
Population: PD Population
Measure: Count of Participants; unit: Participants
Arm/Group | LBP-EC01 | Placebo
Number analyzed (Participants) | 21 | 7
Participants
  Day 2 | 11 | 2
  Day 3 | 8 | 2
  Day 5 | 10 | 4
  Day 7 | 9 | 3
  Day 14 | 8 | 5
  Day 28/ET | 9 | 3

6. Secondary Outcome: Time to 1 Logarithmic Reduction in Urinary E.Coli Count From Baseline
Description: The secondary objective of this study was to evaluate the pharmacodynamics (PD) of LBP-EC01 through time to 1 logarithmic reduction in urinary E.coli count from baseline
Time Frame: 28 days
Population: PD Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LBP-EC01 | Placebo
Number analyzed (Participants) | 21 | 7
days | 5.9 (7.33) | 8.4 (5.41)

7. Secondary Outcome: Recurrence of E.Coli Colonization or Incidence of Infection Based on Clinical Signs and Symptoms
Description: The secondary objective of this study was to evaluate the pharmacodynamics (PD) of LBP-EC01 through recurrence of E.Coli colonization or incidence of infection based on clinical signs and symptoms
Time Frame: 28 days
Population: PD Population
Measure: Count of Participants; unit: Participants
Arm/Group | LBP-EC01 | Placebo
Number analyzed (Participants) | 21 | 7
Participants | 3 | 0

8. Secondary Outcome: Changes in Immunoglobulin (Ig)A
Description: The secondary objective of this study was to evaluate the pharmacodynamics (PD) of LBP-EC01 through changes in IgA
Time Frame: 28 days
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | LBP-EC01 | Placebo
Number analyzed (Participants) | 24 | 12
participants
  Baseline: (Patients with positive detection (>ULN)) | 2 | 0
  Day 28/ET: (Patients with positive detection (>ULN)): number analyzed (Participants) | 24 | 11
  Day 28/ET: (Patients with positive detection (>ULN)) | 2 | 2

9. Secondary Outcome: Changes in IgE
Description: The secondary objective of this study was to evaluate the pharmacodynamics (PD) of LBP-EC01 through changes in IgE with a positive detection of >100 IU/mL
Time Frame: 28 days
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | LBP-EC01 | Placebo
Number analyzed (Participants) | 24 | 12
participants
  Baseline: Patients with positive detection (>ULN) | 7 | 3
  Day 28/ET: Patients with positive detection (>ULN): number analyzed (Participants) | 24 | 11
  Day 28/ET: Patients with positive detection (>ULN) | 8 | 2

10. Secondary Outcome: Changes in IgG
Description: The secondary objective of this study was to evaluate the pharmacodynamics (PD) of LBP-EC01 through changes in IgG with a positive detection of >1600 mg/dL (>16.0 g/L)
Time Frame: 28 days
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | LBP-EC01 | Placebo
Number analyzed (Participants) | 24 | 12
participants
  Baseline: Patients with positive detection (>ULN) | 1 | 0
  Day 28/ET: Patients with positive detection (>ULN): number analyzed (Participants) | 24 | 11
  Day 28/ET: Patients with positive detection (>ULN) | 0 | 1

11. Secondary Outcome: Changes in IgM
Description: The secondary objective of this study was to evaluate the pharmacodynamics (PD) of LBP-EC01 through changes in IgM with a positive detection >230 mg/dL (>2.3 g/L)
Time Frame: 28 days
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | LBP-EC01 | Placebo
Number analyzed (Participants) | 24 | 12
participants
  Baseline: Patients with positive detection (>ULN) | 0 | 1
  Day 28/ET: Patients with positive detection (>ULN) | 0 | 0

ADVERSE EVENTS:
Time Frame: 35 days
Arm/Group | LBP-EC01 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/24 | 1/12
Other Adverse Events (participants affected / at risk) | 18/24 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LBP-EC01 (N=24) | Placebo (N=12)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Coronavirus test positive (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LBP-EC01 (N=24) | Placebo (N=12)
Vomiting (Gastrointestinal disorders) | 2 | 0
Headache (Nervous system disorders) | 5 | 0
Dizziness (Nervous system disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Dysuria (Renal and urinary disorders) | 2 | 0
Hematuria (Renal and urinary disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 0
Bladder discomfort (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Catheter site pain (General disorders) | 0 | 1
Urinary tract infections (Infections and infestations) | 5 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Spleen palpable (Investigations) | 1 | 1
Coronavirus test positive (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT04191148/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT04191148/SAP_001.pdf